CLINICAL TRIAL: NCT01102504
Title: Supplementation of Lycopene on Carotid Atheroma: Neovascularisation and Morphology (SOLANUM) Study
Brief Title: Supplementation of Lycopene in Carotid Atheroma
Acronym: SOLANUM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Karol Palwel Budohoski, Resident in Neurosurgery, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SOLANUM 2.0.0
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Carotid Atherosclerotic Disease
Keywords: carotid atheroma; plaque vulnerability; stroke risk
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tomato extract (Ateronon) (Experimental): Supplementation of tomato extract containing 28 mg/day for 12 months in addition to routine treatment.
  Interventions: Dietary Supplement: Ateronon
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Dietary Supplement: Ateronon — Tomato extract containing 28 mg lycopene/ day
  Arms: Tomato extract (Ateronon)

SUMMARY:
Stroke is the second leading cause of death worldwide. One of the causes of stroke which can be treated is narrowing of the carotid artery. Currently the only definite treatment option is surgery or endovascular treatment. All patients not qualified for or awaiting surgery are, therefore, left with best medical therapy and with a yearly risk of stroke anywhere between 1% - 35% depending on the severity of the disease.

The study will use the properties of a tomato extract containing lycopene. Previously studies have demonstrated beneficial properties of tomato extracts:

1. It decreases lipid oxidation
2. It decreases DNA damage
3. It has properties that reduce the speed and amount of cell divisions that inflammatory and smooth muscle cells undergo (both of these cell types contribute to atheroma formation).

The investigators wish to assess whether long-term food supplementation with a tomato extract containing lycopene could influence atherosclerotic plaque characteristics. The investigators will assess this using Magnetic Resonance Imaging of the plaque and transcranial Doppler ultrasonography for counting the number of blood clots that go to the brain's arteries. Furthermore the investigators wish to examine the effect of long-term food supplementation with a tomato extract containing lycopene on blood cholesterol levels and lipid oxidation and blood markers of inflammation and injury of the inner lining of the arteries.

This will be a single center, double blind, randomised, placebo controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 - 90 years old,
* Clinically documented carotid symptomatic atherosclerotic disease (symptomatic disease will be considered if one of the following has occurred within 2 months prior to symptoms:

  1. Amaurosis fugax
  2. Transient ischemic attack (TIA)
  3. Stroke (ipsilaterally to the stenotic artery)
* >30% stenosis on initial B-mode ultrasonography imaging,
* Written, informed consent.

Exclusion Criteria:

* Age <40 years old or >90 years old,
* Time from symptom to recruitment > 2 months
* <30% stenosis on B-mode ultrasonography imaging,
* Scheduled for surgical/endovascular intervention within 3 months,
* High-dose statin therapy (>80 mg/day fluvastatin; >40 mg/day simvastatin; >40 mg/day pravastatin; >10 mg/day atorvastatin; >10 mg/day rosuvastatin 21),
* Other lipid-lowering therapy (fibric acid derivatives, niacin ≥250 mg/day, resins, ezetimibe, fish-oil supplements),
* Chronic use of high dose aspirin >325 mg/day,
* Allergy or hypersensitivity to tomatoes and tomato products, gadolinium and history of any other significant atopy/allergy (e.g. soy, whey, lutein, lecithin),
* Contraindications for MRI studies including claustrophobia, any MRI non-compatible devices implanted (vascular clips, metal sutures, craniofix, cardiac pacers, endovascular stents/coils, etc.),
* Known renal impairment with creatinine clearance <50 ml/min (as per departmental policy),
* Women of childbearing potential,
* Inability to consent

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2017-12 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Plaque morphology and biomechanics on magnetic resonance | 12 months
  Magnetic resonance imiging (MRI) of the plaques will be performed with detailed assessment of plaque morphological parameters: fibrous cap, lipid rich necrotic core, intraplaque hemorrhage. Sheer stress and wall stress will be calculated using magnetic resonance data.
Serum levels of lycopene - a component of the tomato extract | 12 months
  Serum levels of lycopene obtained through long-time supplementation with a tomato extract containing lycopene.
Microemboli on transcranial Doppler (TCD) | 12 months
  Amount of microeboli detected using bilateral middle cerebral artery (MCA) TCD monitoring (DWL, Germany, 2-MHz probe). TCD will be performed by a single investigator (KPB) for 1 hour

SECONDARY OUTCOMES:
Biochemistry | 12 months
  Serum levels of total cholesterol, low-denisty lipoproteins (LDL), oxidized-LDL (oxy-LDL), high-density lipoproteins (HDL), C-reactive protein (CRP) as biomarkers of atherosclerosis
Levels of blood circulating endothelial cells and endothelial progenitor cells | 12 months
  Levels of blood circulating endothelial cells and endothelial progenitor cells will be measured as markers for endothelial injury
Plaque neovascularisation | 12 months
  Plaque enhancement on dynamic contrast-enhanced MRI perfusion imaging using gadolinium-based contrast agent as a surrogate marker for plaque inflammation and neovascularisation.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan H Gillard, FRCR, Principal Investigator — University Department of Radiology, University of Cambridge, Addenbrooke's Hospital, Hills Road, CB2 0QQ Cambridge, UK
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Background] Corti R, Fuster V, Fayad ZA, Worthley SG, Helft G, Smith D, Weinberger J, Wentzel J, Mizsei G, Mercuri M, Badimon JJ. Lipid lowering by simvastatin induces regression of human atherosclerotic lesions: two years' follow-up by high-resolution noninvasive magnetic resonance imaging. Circulation. 2002 Dec 3;106(23):2884-7. doi: 10.1161/01.cir.0000041255.88750.f0. PMID 12460866
- [Background] Corti R, Fuster V, Fayad ZA, Worthley SG, Helft G, Chaplin WF, Muntwyler J, Viles-Gonzalez JF, Weinberger J, Smith DA, Mizsei G, Badimon JJ. Effects of aggressive versus conventional lipid-lowering therapy by simvastatin on human atherosclerotic lesions: a prospective, randomized, double-blind trial with high-resolution magnetic resonance imaging. J Am Coll Cardiol. 2005 Jul 5;46(1):106-12. doi: 10.1016/j.jacc.2005.03.054. PMID 15992643
- [Background] Tang TY, Howarth SP, Miller SR, Graves MJ, Patterson AJ, U-King-Im JM, Li ZY, Walsh SR, Brown AP, Kirkpatrick PJ, Warburton EA, Hayes PD, Varty K, Boyle JR, Gaunt ME, Zalewski A, Gillard JH. The ATHEROMA (Atorvastatin Therapy: Effects on Reduction of Macrophage Activity) Study. Evaluation using ultrasmall superparamagnetic iron oxide-enhanced magnetic resonance imaging in carotid disease. J Am Coll Cardiol. 2009 Jun 2;53(22):2039-50. doi: 10.1016/j.jacc.2009.03.018. PMID 19477353
- [Background] Underhill HR, Yuan C, Zhao XQ, Kraiss LW, Parker DL, Saam T, Chu B, Takaya N, Liu F, Polissar NL, Neradilek B, Raichlen JS, Cain VA, Waterton JC, Hamar W, Hatsukami TS. Effect of rosuvastatin therapy on carotid plaque morphology and composition in moderately hypercholesterolemic patients: a high-resolution magnetic resonance imaging trial. Am Heart J. 2008 Mar;155(3):584.e1-8. doi: 10.1016/j.ahj.2007.11.018. Epub 2008 Jan 18. PMID 18294500
- [Background] Carpenter KL, Hardwick SJ, Albarani V, Mitchinson MJ. Carotenoids inhibit DNA synthesis in human aortic smooth muscle cells. FEBS Lett. 1999 Mar 19;447(1):17-20. doi: 10.1016/s0014-5793(99)00252-5. PMID 10218573
- [Background] Das S, Otani H, Maulik N, Das DK. Lycopene, tomatoes, and coronary heart disease. Free Radic Res. 2005 Apr;39(4):449-55. doi: 10.1080/10715760500053685. PMID 16032783
- [Background] Holvoet P, Collen D. Oxidation of low density lipoproteins in the pathogenesis of atherosclerosis. Atherosclerosis. 1998 Apr;137 Suppl:S33-8. doi: 10.1016/s0021-9150(97)00305-5. PMID 9694539